CLINICAL TRIAL: NCT03704259
Title: Nano-Ceramic Coating for Laparoscope Lens: a Cheap Magical Solution for Lens Fogging and Smearing
Brief Title: Nano-Ceramic Coating for Laparoscope Lens
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, yousef ahmed el-ayman, Dr., Master's degree, assistant lecturer of general surgery, Zagazig University
Other Study IDs: ZagazigELSU
Record Dates: First submitted 2018-09-12; First posted 2018-10-12 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Laparoscopic Surgical Procedures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Other: Ceramic coating — coating the laparoscope lens with commercial brand ceramic coating, bought from car service centers specialized in such applications
  Other Names: nan-ceramic coating

SUMMARY:
The investigator tests the effectiveness of nano-ceramic coating when applied (painted) on laparoscope lens to protect it from fogging or smearing during laparoscopic operations

DETAILED DESCRIPTION:
A Ceramic Coating is a liquid polymer that is applied by hand to surfaces to make them resistant to scratching, staining, rust or oxidation, as well as "hydrophilic", meaning that water or mud doesn't stick to them and so, they become much easier to clean. It was publicly commercialized in recent years for use on automobiles to preserve their gloss, protect their paint, preserve the clarity of their wind shields and headlights so as to provide better lighting and vision.

On the other hand, lens fogging and other vision-obstructing events during laparoscopic or endoscopic operations(e.g. being smeared by blood or other body fluids during operation, or having a piece of loose tissue stick to its surface that require manual removal and wiping) have been an ever-lasting concern for operators ever since the advent of the respective devices. Many techniques and methods have developed, tested and compared regarding their effectiveness in protecting the lens from such events and preserving vision clear and uninterrupted during operations. Examples of such methods are (scope warmers, FREDTM, ResoclearTM, chlorhexidine, betadine and immersion in heated saline.

In this study the investigator seeks to apply the idea of nano-ceramic coating as a new technique for achieving that goal. to the investigator's best knowledge, this idea was never conceived or tested in the field before.

ELIGIBILITY:
Inclusion Criteria:

* Any patient requiring laparoscopic operation

Exclusion Criteria:

* Any intra-operative event or obstacle that requires conversion to open surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted for laparoscopic operations
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
rate of fogging or smearing (per hour) | One month
  The investigator calculates the number of times the lens is visibly fogged or smeared per hour of operation.
rate of fogging or smearing (per single operation) | One month
  The investigator calculates the number of times the lens is visibly fogged or smeared during a single operation.
rate of extraction for cleaning (per hour) | One month
  The investigator calculates the number of times the lens needs to be extracted from the abdomen for cleaning per hour of operation.
Rate of extraction for cleaning (per operation) | One month
  The investigator calculates the number of times the lens needs to be extracted from the abdomen for cleaning per single operation.
The time consumption for lens cleaning (per hour) | One month
  The investigator calculates the time consumption of the cleaning process as a total (in minutes) per hour.
The time consumption for lens cleaning (per single operation) | One month
  The investigator calculates the time consumption of the cleaning process as a total (in minutes) per single operation.
Cleaning difficulty (per hour) | One month
  The investigator calculates how many times the lens needed more measures for cleaning than simple wiping E.G immersion in hot saline per hour
Cleaning difficulty (per single operation) | One month
  The investigator calculates how many times the lens needed more measures for cleaning than simple wiping E.G immersion in hot saline per hour

SECONDARY OUTCOMES:
Affecting the lens function | One month
  This is a subjective assessment measure, represented by the operators' statement about whether coating the lens affected its vision I.E whether there is a difference in acuity of vision between the coated and the non-coated lens in the absence of any fogging or smearing.
  Statement is given as one of five choices:
  1. coated lens is notably better (significant difference)
  2. coated lens is slightly better (negligible difference)
  3. non-coated lens is notably better (significant difference)
  4. non-coated lens is slightly better (negligible difference)
  5. no difference

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University, Zagazig, Elsharkia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manning TG, Papa N, Perera M, McGrath S, Christidis D, Khan M, O'Beirne R, Campbell N, Bolton D, Lawrentschuk N. Laparoscopic lens fogging: solving a common surgical problem in standard and robotic laparoscopes via a scientific model. Surg Endosc. 2018 Mar;32(3):1600-1606. doi: 10.1007/s00464-017-5772-x. Epub 2017 Aug 8. PMID 28791559